CLINICAL TRIAL: NCT03679143
Title: A Phase 1 Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ZSP1273 and the Effect of Food on ZSP1273 Pharmacokinetics in Chinese Healthy Subjects.
Brief Title: The Safety, Tolerability and Pharmacokinetic Study of ZSP1273 in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Zhongsheng Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZSP1273-18-01
Record Dates: First submitted 2018-09-18; First posted 2018-09-20 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — ZSP1273

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking for Participant, Investigator and Clinical Research Associate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- ZSP1273(single dose)-100 mg(Cohort 1) (Experimental): ZSP1273 100 mg /Placebo
  Interventions: Drug: ZSP1273 100 mg; Drug: Placebo 100 mg
- ZSP1273(single dose)-200 mg(Cohort 2) (Experimental): ZSP1273 200mg/Placebo
  Enrollment into Cohort 2 will begin upon assurance of tolerance for Cohort 1.
  Interventions: Drug: ZSP1273 200 mg; Drug: Placebo 200 mg
- ZSP1273(single dose)-400 mg(Cohort 3) (Experimental): ZSP1273 400mg/Placebo
  Enrollment into Cohort 3 will begin upon assurance of tolerance for Cohort 2.
  Interventions: Drug: ZSP1273 400 mg; Drug: Placebo 400 mg
- ZSP1273(single dose)-600 mg(Cohort 4) (Experimental): ZSP1273 600 mg/Placebo
  Enrollment into Cohort 4 will begin upon assurance of tolerance for Cohort 3.
  Interventions: Drug: ZSP1273 600 mg; Drug: Placebo 600 mg
- ZSP1273(single dose)-900 mg(Cohort 5) (Experimental): Drug:ZSP1273 900 mg/Placebo 900mg；
  Enrollment into Cohort 5 will begin upon assurance of tolerance for Cohort 4.
  Interventions: Drug: ZSP1273 900 mg; Drug: Placebo 900 mg
- ZSP1273(single dose)-1200 mg(Cohort 6) (Experimental): ZSP1273 1200 mg/Placebo
  Enrollment into Cohort 6 will begin upon assurance of tolerance for Cohort 5.
  Interventions: Drug: ZSP1273 1200 mg; Drug: Placebo 1200 mg
- ZSP1273(Food Effect)-Cohort 7 (Experimental): Drug:ZSP1273 /Placebo； Period 1 (Day1 to Day5): Subjects receive ZSP1273/Placebo under the fasting or fed condition ,respectively on Day1.
  Period 2 (Day 8 to Day12): Subjects receive ZSP1273/Placebo under the fed or fasting condition, respectively on Day 8.
  Interventions: Drug: ZSP1273; Drug: Placebo
- ZSP1273(multiple doses)-Low Dose(Cohort 8) (Experimental): while fasted or fed according to the results of Cohort FE
  ZSP1273 /Placebo for 5 Days.
  Interventions: Drug: ZSP1273 Low Dose; Drug: Placebo
- ZSP1273(multiple doses)-Median Dose(Cohort 9) (Experimental): while fasted or fed according to the results of Cohort FE
  ZSP1273/Placebo for 5 Days.
  Interventions: Drug: ZSP1273 Median Dose; Drug: Placebo
- ZSP1273(multiple doses)-High Dose(Cohort 10) (Experimental): while fasted or fed according to the results of Cohort FE
  ZSP1273/Placebo for 5 Days.
  Interventions: Drug: ZSP1273 High Dose; Drug: Placebo

INTERVENTIONS:
Drug: ZSP1273 100 mg — ZSP1273 tablet administered orally once daily under fasted condition
  Arms: ZSP1273(single dose)-100 mg(Cohort 1)
Drug: Placebo 100 mg — Participants will receive placebo matching to ZSP1273 orally once daily in the fasting state.
  Arms: ZSP1273(single dose)-100 mg(Cohort 1)
Drug: ZSP1273 200 mg — ZSP1273 tablets administered orally once daily under fasted condition
  Arms: ZSP1273(single dose)-200 mg(Cohort 2)
Drug: Placebo 200 mg — Participants will receive placebo matching to ZSP1273 orally once daily under fasted condition
  Arms: ZSP1273(single dose)-200 mg(Cohort 2)
Drug: ZSP1273 400 mg — ZSP1273 tablets administered orally once daily in the fasting state
  Arms: ZSP1273(single dose)-400 mg(Cohort 3)
Drug: Placebo 400 mg — Participants will receive placebo matching to ZSP1273 orally once daily in the fasting state
  Arms: ZSP1273(single dose)-400 mg(Cohort 3)
Drug: ZSP1273 600 mg — ZSP1273 tablets administered orally once daily under fasted condition
  Arms: ZSP1273(single dose)-600 mg(Cohort 4)
Drug: Placebo 600 mg — Participants will receive placebo matching to ZSP1273 orally once daily under fasted condition
  Arms: ZSP1273(single dose)-600 mg(Cohort 4)
Drug: ZSP1273 900 mg — ZSP1273 tablets administered orally once daily in the fasting state
  Arms: ZSP1273(single dose)-900 mg(Cohort 5)
Drug: Placebo 900 mg — Participants will receive placebo matching to ZSP1273 orally once daily under fasted condition
  Arms: ZSP1273(single dose)-900 mg(Cohort 5)
Drug: ZSP1273 1200 mg — ZSP1273 tablets administered orally once daily in the fasting state
  Arms: ZSP1273(single dose)-1200 mg(Cohort 6)
Drug: Placebo 1200 mg — Participants will receive placebo matching to ZSP1273 orally once daily in the fasting state
  Arms: ZSP1273(single dose)-1200 mg(Cohort 6)
Drug: ZSP1273 — ZSP1273 tablets administered orally once daily under fasted or fed condition
  Arms: ZSP1273(Food Effect)-Cohort 7
Drug: Placebo — Participants will receive placebo matching to ZSP1273 orally once daily under fasted or fed condition
  Arms: ZSP1273(Food Effect)-Cohort 7
Drug: ZSP1273 Low Dose — ZSP1273 tablets administered orally once daily under fasted or fed condition for 5 Days.
  Arms: ZSP1273(multiple doses)-Low Dose(Cohort 8)
Drug: Placebo — Participants will receive placebo matching to ZSP1273 orally once daily under fasted or fed condition for 5 Days.
  Arms: ZSP1273(multiple doses)-Low Dose(Cohort 8)
Drug: ZSP1273 Median Dose — ZSP1273 tablets administered orally twice daily for 4 Days and once daily on Day 5 under fasted or fed condition.
  Arms: ZSP1273(multiple doses)-Median Dose(Cohort 9)
Drug: Placebo — Participants will receive placebo matching to ZSP1273 orally twice daily for 4 Days and once daily on Day 5 under fasted or fed condition.
  Arms: ZSP1273(multiple doses)-Median Dose(Cohort 9)
Drug: ZSP1273 High Dose — ZSP1273 tablets administered orally twice daily for 4 Days and once daily on Day 5 under fasted or fed condition.
  Arms: ZSP1273(multiple doses)-High Dose(Cohort 10)
Drug: Placebo — Participants will receive placebo matching to ZSP1273 orally twice daily for 4 Days and once daily on Day 5 under fasted or fed condition.
  Arms: ZSP1273(multiple doses)-High Dose(Cohort 10)

SUMMARY:
This is a single center,double-blind,randomized,parallel design, single and multiple dose trial to evaluate the pharmacokinetics(PK), safety and tolerability of ZSP1273,and the effect of food on ZSP1273 Pharmacokinetics.

DETAILED DESCRIPTION:
The study will be divided in 3 parts :

Study Part I(Single Ascending Dosing, SAD) will be a single ascending dose to be run at a maximum of 6 dose levels. Subjects included in this part of the study will receive only one dose level to limit the exposure to ZSP1273. Four subjects are planned to be included in the first group while 10 subjects are enrolled in every following cohort.

Study Part II(Multiple Ascending Dosing, MAD) will start after completion of some Cohorts of Study Part I. Study Part II will be a multiple ascending dose to be run at a maximum of 3 dose levels. Subjects included in this part of the study will receive only one dose level. This part also enrolls 10 subjects in every cohort.

Study Part III(Food Effect study, FE) will consists of 2 periods,and subjects will receive a single dose ranged from 100-600mg on fasting and postprandial states respectively. There will be a 7-day wash out period between treatment periods.A total of 12 to 18 subjects will be included.

All the 3 parts will be run in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

Subjects are required to meet the following criteria in order to be included in the trial:

1. Signature of a dated Informed Consent Form (ICF) indicating that the subject has been informed of all the relevant aspects(including adverse events) of the trial prior to enrollment.
2. Subjects must be willing and able to adhere to the visit schedule and protocol requirements and be available to complete the study.
3. Subjects (including partners) must use reliable methods of contraception during the study and until 6 months following the last dose of investigational product.
4. Males and female subjects between 18-50 years (Both inclusive).
5. Body weight is no less than 50 kg in males and no less than 45 kg in females. Body mass index (BMI) 18≤BMI≤28 kg/m2; BMI is determined by the following equation: BMI = weight/height2 (kg/m2).
6. Physical condition and vital signs: Normal or abnormality has no clinical significance.

Exclusion Criteria:

Eligible subjects must not meet any of the following exclusion criteria:

1. Known hypersensitivity and/or allergy to some drugs and food, especially for the composition that is similar to the investigative product;
2. The average daily smoking are more than 5 cigarettes within 3 months prior to screening.
3. Known history of drug or alcohol abuse.(defined as consumption of 14 units of alcohol per week: 1 unit = 285 ml of beer; or the equivalent of 25 ml of spirit, or 100 ml of wine )
4. Subjects who donated blood or bleeding profusely (> 400 mL) in the 3 months preceding study screening.
5. Dysphagia or any medical history in gastrointestinal that interferes with the absorption of drugs, include a history of frequent nausea or vomit causes by any etiology.
6. History or presence of any disease or condition known to increase the risk of bleeding , eg. acute gastritis, duodenal ulcer, etc.
7. Participant with any history of clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, or urticaria.
8. Subjects with recent significant change in diet or exercise.
9. Participated in another clinical research study and received any investigational products within 3 months prior to dosing.
10. Concomitant therapy with any drugs with known hepatic enzyme-inducing or inhibiting agents prior to screening or during the study, including strong inhibitory agents and inducers that affect metabolic enzymes (see appendix 6 for specific drug information).
11. Use of any prescription or over-the-counter (OTC) medications, vitamins and herbal or dietary supplements within 14 days prior to screening.
12. History of having any special food (including dragon fruit, mango, grapefruit, etc.), strenuous exercises, or other factors may interfere with the absorption, distribution, metabolism, or excretion of drug within 14 days prior to screening.
13. Inability to consume the food provided in the study ( a high fat, high calorie meal includes two eggs , a piece of butter bacon toast, a box of fried potatoes, and a glass of whole milk).This requirement only applies to subjects under fed condition.
14. Presence of clinically significant abnormalities in ECG or QTcB>470ms in males, or QTcB>480ms in females.
15. Pregnancy or breastfeeding at screening and during the study. All female subjects of childbearing potential must have a negative urine pregnancy test at screening and during the trial.
16. Any clinically significant abnormality upon physical examination or presence of a clinically significant gastrointestinal, renal, hepatic, neurologic, hematic, endocrine, neoplastic, pulmonary, immune, psychiatric or cardiovascular and cerebrovascular disorder(s)(but not limited to above disorders) in the 6 months preceding study screening.
17. Positive hepatitis B surface antigen, hepatitis C virus antibody,human immunodeficiency virus (HIV) or treponema pallidum antibodies at screening.
18. Any acute illness or concomitant medication from screening to first dosing.
19. Have chocolate, any food or beverage that contains caffeine or xanthine within 24 hours prior to dosing.
20. Positive for urine drug screening or history of substance and drug abuse for a period of 5 consecutive years before screening.
21. Subjects who may not complete the study for other reasons or should not be included in the study in the opinion of the investigator.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Number and severity of treatment-emergent adverse events (TEAEs) and Serious Adverse Events(SAE) | At day 5, 9, 12 days post first dosing for SAD, MAD, FE part respectively
  Number of participants with TEAEs as assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
Tmax | UP to 5, 9, 12 days for SAD, MAD, FE part respectively
  The time after dosing when Cmax occurs (Tmax)
Cmax | UP to 5, 9, 12 days for SAD, MAD, FE part respectively
  Maximum concentration (Cmax)
t1/2z | UP to 5, 9, 12 days for SAD, MAD, FE part respectively
  t1/2z is defined as the time to decline half of the drug concentration in plasma.
AUCinf（AUC0-∞） | UP to 5, 9, 12 days for SAD, MAD, FE part respectively
  Area under the curve extrapolated until time is infinity (AUCinf)
AUClast（AUC0-t） | UP to 5, 9, 12 days for SAD, MAD, FE part respectively
  AUClast is defined as the concentration of drug from time zero to the last quantifiable concentration.
CL/F | UP to 5, 9, 12 days for SAD, MAD, FE part respectively
  CL/F is defined as the ratio of total clearance(Cl) to bioavailability(F).
λz | UP to 5, 9, 12 days for SAD, MAD, FE part respectively
  λz is defined as the ratio between the elimination of compound per unit time and the total amount of compound.
CLr | UP to 5, 9, 12 days for SAD, MAD, FE part respectively
  CLr is defined as how many milliliters of plasma in which some substance can be completely eliminated in the unit time (per minute) of two kidneys.
Food Effect PK Parameter: Fe0-t | UP to 12 days
  Fe0-t is defined as the cumulative excretion rate of the drug in urine and feces.
Food Effect PK Parameter: Ae | UP to 12 days
  Ae is defined as the amount of unchanged drug excreted in urine or faeces after administration.
Multiple-dose plasma PK parameter: Rac of ZSP1273 at steady state | Up to 9 days
  Rac (Accumulation Index) is defined as the ratio between AUC0-XX in Day XX and AUC0-XX in Day1
Multiple-dose plasma PK parameter: DF of ZSP1273 at steady state | Up to 9 days
  DF is defined as the percentage of fluctuation in steady state is 100 * (Cmax, ss - Cmin, ss)/Cavg, ss.
Multiple-dose plasma PK parameter: Cmin of ZSP1273 at steady state | Up to 9 days
  Cmin is defined as the minimum observed concentration of drug in plasma at steady state.

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, MD, Principal Investigator — The First Hospital of Jilin University; Shucheng Hua, MD, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Derived] Hu Y, Li H, Wu M, Zhang H, Ding Y, Peng Y, Li X, Yu Z. Single and multiple dose pharmacokinetics and safety of ZSP1273, an RNA polymerase PB2 protein inhibitor of the influenza A virus: a phase 1 double-blind study in healthy subjects. Expert Opin Investig Drugs. 2021 Nov;30(11):1159-1167. doi: 10.1080/13543784.2021.1994944. Epub 2021 Nov 1. PMID 34654349